CLINICAL TRIAL: NCT04752358
Title: A Phase 2 Open-Label Clinical Trial of ADP-A2M4CD8 in Subjects With Advanced Esophageal or Esophagogastric Junction Cancers
Brief Title: ADP-A2M4CD8 in HLA-A2+ Subjects With MAGE-A4 Positive Esophageal or Esophagogastric Junction Cancers (SURPASS-2)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated due to difficulty recruiting subjects and lack of efficacy
Sponsor: Adaptimmune (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADP-0055-002
Record Dates: First submitted 2021-02-08; First posted 2021-02-12 (Actual); Results first posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-08

CONDITIONS: Esophageal Cancer; Esophagogastric Junction Cancer
Keywords: Cell Therapy; T Cell Therapy; SPEAR T Cell; MAGE-A4; Immuno-oncology; Metastatic; Esophagogastric Junction; Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous genetically modified ADP-A2M4CD8 cells (Experimental)
  Interventions: Genetic: Autologous genetically modified ADP-A2M4CD8 cells

INTERVENTIONS:
Genetic: Autologous genetically modified ADP-A2M4CD8 cells — Infusion of autologous genetically modified ADP-A2M4CD8 on Day 1

SUMMARY:
This study will investigate the efficacy of ADP-A2M4CD8 T-cell therapy in subjects who have the appropriate human leukocyte antigen (HLA) and tumor antigen status and whose esophageal or esophagogastric junction (EGJ) cancer expresses the MAGE-A4 protein.

ELIGIBILITY:
Key Inclusion Criteria:

* Age ≥18 and <75 years
* Diagnosis of Esophageal cancer or Esophagogastric junction cancer.
* Previously received treatment for advanced or metastatic disease.
* Measurable disease according to RECIST v1.1.
* HLA-A*02 positive
* Tumor shows MAGE-A4 expression confirmed by central laboratory.
* ECOG Performance Status of 0 or1.
* Left ventricular ejection fraction (LVEF) ≥50%.

Note: other protocol defined Inclusion criteria may apply

Key exclusion criteria

1. Positive for any HLA-A*02 allele other than: one of the inclusion alleles
2. History of allergic reactions attributed to compounds of similar chemical or biologic composition to fludarabine, cyclophosphamide or other agents used in the study
3. Active autoimmune or immune mediated disease
4. Leptomeningeal disease, carcinomatous meningitis or symptomatic CNS metastases
5. Other prior malignancy that is not considered by the Investigator to be in complete remission. Clinically significant cardiovascular disease
6. Uncontrolled intercurrent illness
7. Active infection with human immunodeficiency virus, hepatitis B virus, hepatitis C virus, or human T cell leukemia virus
8. Pregnant or breastfeeding

Note: other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-06-09 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - University of Chicago Medicine, Chicago, Illinois
  - Washington University School of Medicine- Siteman Cancer Center, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - University Of Texas, MD Anderson Cancer Center, Houston, Texas
  - University Of Wisconsin Clinical Science Center, Madison, Wisconsin
- Canada (2):
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre Glen Site, Montreal, Quebec
- Spain (7):
  - Hospital Universitari Vall d'Hebron, la Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Córdoba, Madrid
  - Hospital Clinico Universitario de Valencia, Ibáñez, Valencia
  - Hospital Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Madrid Sanchinarro (CIOCC), Madrid
  - Clinica Universidad de Navarra, Navarro
  - Hospital Universitario Virgen del Rocio, Seville

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 2 open-label, single treatment, clinical trial of ADP-A2M4CD8 in participants with advanced esophageal or esophagogastric junction cancers
Pre-assignment Details: All participants were assigned to one treatment (ADP-A2M4CD8)
Groups:
- Esophageal: Eligible participants with esophageal cancer who received ADP-A2M4CD8 as a single infusion
- Esophagogastric Junction: Eligible participants with esophagogastric junction cancer who received ADP-A2M4CD8 as a single infusion
Period: Overall Study
Arm/Group | Esophageal | Esophagogastric Junction
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: Eligible participants who received ADP-A2M4CD8 as a single infusion
Groups:
- Total: Total of all reporting groups
Arm/Group | Esophageal | Esophagogastric Junction | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 2 | 1 | 3
Age, Continuous [Median (Full Range); unit: years] | 68 [67 to 69] | 72 [72 to 72] | 69 [67 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) by Independent Radiological Assessment Committee (IRAC)
Description: Confirmed tumor response (complete response [CR] or partial response [PR]) to treatment as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by IRAC
Time Frame: From T-cell infusion to end of Interventional Phase (Up to 5 months from T-cell infusion).
Population: Participants who received ADP-A2M4CD8. No subject images were assessed by Independent Reviewer due to lack of efficacy observed on Investigator review. Thus, no results are reported.
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number and Percentage of Participants With Adverse Events (AEs) Including Serious Adverse Events (SAEs), and Adverse Events of Special Interest (AESI)
Description: An AE was defined as any untoward medical occurrence in a subject or clinical study participant temporally associated with the use of the study intervention, whether or not considered related to the study intervention. Therefore, an AE could have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. The number of participants with AEs (including SAEs), SAEs and AESI including cytokine release syndrome, ICANS, and prolonged cytopenia are presented.
Time Frame: From start of lymphodepleting chemotherapy to end of Interventional Phase (up to 5 months)
Population: Participants who received ADP-A2M4CD8
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 2 | 1
Participants
  AE | 2 | 1
  SAE | 1 | 1
  AESI - cytokine release syndrome | 1 | 1
  AESI- ICANS | 0 | 0
  AESI- Prolonged cytopenia | 0 | 1

3. Secondary Outcome: Time to Response (TTR) by IRAC
Description: TTR (CR or PR) was defined as the interval between the date of first T-cell infusion and the earliest date of first documented confirmed CR or confirmed PR.
Time Frame: From T-cell infusion until first documented confirmed CR or PR
Population: Participants who received ADP-A2M4CD8 and had a confirmed CR or PR. No subjects had a confirmed CR or PR. Thus, no results are reported.
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Response (DoR) by IRAC
Description: DoR is defined as duration between the initial date of the confirmed complete or partial response to the date of progressive disease or death, where tumor response and disease progression were assessed by IRAC.
Time Frame: From initial date of first confirmed response (CR or PR) until PD or death
Population: as for outcome 3
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Best Overall Response (BOR) by IRAC
Description: BOR is the best response recorded from the start of T-cell infusion until disease progression as assessed by IRAC. Response categories are confirmed CR, confirmed PR, stable disease (SD) and confirmed progressive disease (PD).
Time Frame: From T-cell infusion until disease progression
Population: as for outcome 1
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Progression Free Survival (PFS) by IRAC
Description: PFS is defined as time from the T-cell infusion to the date of the first documentation of progressive disease (PD) as assessed by IRAC or death due to any cause, whichever occurs first.
Time Frame: From T-cell infusion until first documented PD, as assessed by IRAC, or death due to any cause, whichever occurs first
Population: Participants who received ADP-A2M4CD8. No subject images were assessed by IRAC due to lack of efficacy observed on Investigator review. Hence, no results are reported.
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Overall Response Rate (ORR) by Investigator Assessment
Description: Confirmed tumor response (complete response [CR] or partial response [PR]) to treatment as assessed using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator Assessment
Time Frame: From T-cell infusion to end of Interventional Phase (Up to 5 months from T-cell infusion).
Population: Participants who received ADP-A2M4CD8.
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 2 | 1
Participants | 0 | 0

8. Secondary Outcome: Time to Response (TTR) by Investigator Assessment
Description: as for outcome 3
Time Frame: From T-cell infusion until first documented confirmed CR or PR
Population: Participants who received ADP-A2M4CD8 and had a confirmed CR or PR. No subjects had a confirmed CR or PR. Thus, TTR was not calculated, and no results are reported.
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Duration of Response (DoR) by Investigator Assessment
Description: DoR is defined as duration between the initial date of the confirmed complete or partial response to the date of progressive disease or death, where tumor response and disease progression were assessed by Investigator Assessment.
Time Frame: From initial date of first confirmed response (CR or PR) until PD or death
Population: Participants who received ADP-A2M4CD8 and had a confirmed CR or PR. No subjects had a confirmed CR or PR. Thus, DoR was not calculated, and no results are reported.
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Best Overall Response (BOR) by Investigator Assessment
Description: BOR is the best response recorded from the start of T-cell infusion until disease progression as assessed by the Investigator. Response categories are confirmed CR, confirmed PR, stable disease (SD) and confirmed progressive disease (PD).
Time Frame: From T-cell infusion until disease progression (Up to 5 months)
Population: Participants who received ADP-A2M4CD8.
Measure: Count of Participants; unit: Participants
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 2 | 1
Participants
  Complete Response | 0 | 0
  Partial Response | 0 | 0
  Stable Disease | 2 | 1
  Progressive Disease | 0 | 0

11. Secondary Outcome: Progression Free Survival (PFS) by Investigator Assessment
Description: PFS is defined as the time from the T-cell infusion to the date of the first documentation of progressive disease (PD) as assessed by investigator assessment or death due to any cause, whichever occurs first.
Time Frame: From T-cell infusion until first documented PD, as assessed by Investigator, or death due to any cause, whichever occurs first (up to 5 months)
Population: Participants who received ADP-A2M4CD8
Measure: Median (Full Range); unit: Weeks
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 2 | 1
Weeks | 14.43 [8.14 to 20.71] | 8.43 [8.43 to 8.43]

12. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of first T-cell infusion to the date of death (due to any cause).
Time Frame: From T-cell infusion to death due to any reason (up to 7 months)
Population: Participants who received ADP-A2M4CD8
Measure: Median (Full Range); unit: Weeks
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 2 | 1
Weeks | 19.64 [18.57 to 20.71] | 29.71 [29.71 to 29.71]

13. Secondary Outcome: Replication Competent Lentivirus
Description: The presence of RCL was assessed by qPCR targeting a segment of the vesicular stomatitis virus glycoprotein (VSV G) coding sequence. 1 participant had at least 1 post-infusion sample tested for RCL.
  The count of participants with RCL post-infusion is presented.
Time Frame: From T-cell infusion to end study (up to 7 months)
Population: Participants who received ADP-A2M4CD8 and had a post-infusion sample tested for VSV-G
Measure: Count of Participants; unit: Participants
Groups:
- Esophageal: Eligible participants with esophageal cancer who received ADP-A2M4CD8 as a single infusion and a post-infusion sample tested for VSV-G (RCL)
- Esophagogastric Junction: Eligible participants with esophagogastric junction cancer who received ADP-A2M4CD8 as a single infusion and a post-infusion sample tested for VSV-G (RCL)
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 1
Participants | 0 | 0

14. Secondary Outcome: Insertional Oncogenesis (IO)
Description: Deoxyribonucleic acid (DNA) from participants peripheral blood mononuclear cell (PBMC) samples are subjected to lentiviral vector integration site analysis by next-generation sequencing, thus evaluating both the clonality status of the transduced cell population and the genomic localization of individual integration sites. The outcome measure is the number of participants with integration sites representing more than 5% of all unique sites.
Time Frame: From 1 year post T-cell infusion
Population: Participants who received ADP-A2M4CD8 and had a sample analyzed for IO. All subjects died prior to 1 year post T-cell infusion, subsequently no samples were obtained or analyzed.
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 0 | 0

15. Secondary Outcome: Peak Persistence
Description: Peak persistence of ADP-A2M4CD8 cells was reported as vector copy numbers per microgram of genomic DNA from peripheral blood mononuclear cell (PBMC).
Time Frame: From T-cell infusion to end study (up to 7 months)
Population: Participants who received ADP-A2M4CD8
Measure: Median (Full Range); unit: copies/microgram DNA
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 2 | 1
copies/microgram DNA | 59546.3 [41432.7 to 77660] | 135581.5 [135581.5 to 135581.5]

16. Secondary Outcome: Time to Peak Persistence
Description: Time from ADP-A2M4CD8 T-cell infusion to peak persistence of cells.
Time Frame: From T-cell infusion to end study (up to 7 months)
Population: Participants who received ADP-A2M4CD8
Measure: Median (Full Range); unit: Days
Arm/Group | Esophageal | Esophagogastric Junction
Number analyzed (Participants) | 2 | 1
Days | 11.5 [8 to 15] | 17 [17 to 17]

17. Secondary Outcome: Concordance of the MAGE A-4 Clinical Trial Assay and in Vitro Diagnostic (IVD) Kit.
Description: Concordance of the MAGE A-4 clinical trial assay and in vitro diagnostic (IVD) kit.
Time Frame: Screening visit
Population: Due to study termination, an IVD kit for companion diagnosis was not developed. Thus, there is no data to report regarding concordance of the MAGE A-4 clinical trial assay and the IVD companion diagnostic kit.
Groups:
- All Screened Participants: All participants who were screened and had slides available for MAGE A4 assay
Arm/Group | All Screened Participants
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from the start of lymphodepleting chemotherapy until the end of the interventional phase (up to 5 months). Deaths were collected from start of lymphodepletion chemotherapy until the end of the study (up to 7 months).
Description: Serious adverse events were reported for all participants who received ADP-A2M4CD8
Arm/Group | Esophageal | Esophagogastric Junction
All-Cause Mortality (participants affected / at risk) | 2/2 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esophageal (N=2) | Esophagogastric Junction (N=1)
Cytokine release syndrome (Immune system disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esophageal (N=2) | Esophagogastric Junction (N=1)
Vomiting (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 0 | 1
Migraine with aura (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 1 | 0
Cytomegalovirus infection reactivation (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-11-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT04752358/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-23): https://cdn.clinicaltrials.gov/large-docs/58/NCT04752358/SAP_001.pdf